CLINICAL TRIAL: NCT01905488
Title: Perioperative Changes of Cognitive Function According to Jugular Vein Insufficiency in Robot-assisted Prostatectomy
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2009-0056
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group N: patients who didn't show internal jugula vein valve incompetency (IJVVI)
- Group PT: patients who showed IJVVI after pneumoperitoneum or Trendelenburg position
- Group S: patients who showed IJVVI in supine position

SUMMARY:
Internal jugular vein (IJV) is the main pathway of cerebral venous drainage and it has valve system to prevent retrograde blood flow to the brain. Anatomical studies revealed that bicuspid or tricuspid valves were located in both jugular veins 2 cm above the subclavia-jugulars bifurcation and 7-18% of the valves were incompetent. IJVV incompetence (IJVVI) may result in retrograde flow which leads to brain congestion and increase of intracranial pressure, which can cause brain dysfunctions in some patients. IJVVI has been reported to be associated with transient global amnesia (TGA), cough syncope, exertional headache, transient ischemic attack, and air embolism. Demographic data are associated with the development of IJVVI. Akkawi et al. demonstrated that old age over 50 years and male gender are the risk factors for IJVVI. A few physiologic conditions are related with IJVVI including elevated intra-thoracic and intra-abdominal pressure, and pulmonary hypertension. Robot assisted laparoscopic prostatectomy (RLP) is one of the most common robotic surgery because of its significant benefits such as smaller incision, less severe postoperative pain, less intraoperative bleeding, and shorter hospital stay compared to traditional radical prostatectomy. The patients undergoing RLP are mostly over 60 years old, have neurologic, cardiac and pulmonary comorbidities. For RLP, patients are in Trendelenburg position most of the time during surgery, which could cause increases in intra-abdominal and intrathoracic pressure.

ELIGIBILITY:
Inclusion Criteria:

* over 50 years old
* ASA class I or II
* Scheduled for robot assisted laparoscopic prostatectomy

Exclusion Criteria:

* previous neurologic deficit
* history of psychiatric disease, alcoholism or other drug dependency
* Serious hearing or visual impairment or any other comorbidities which would preclude neuropsychological tests

Ages: 56 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were over 50 years old with ASA class I or II, scheduled for robot-assisted laparoscopic prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change of neurocognitive function from baseline at 2 days after surgery | 2 days after surgery
  Six neurocognitive function tests( 1. Mini-Mental State Examination 2. Auditory Verbal Learning Test 3. Digit Symbol Substitution Test 4. Color Word Stroop Test 5. Digit Span Test 6. Grooved Pegboard Test ) were performed 1 day before surgery as a baseline, then 2 days after surgery as primary outcome parameters. The values between 2 observations were compared to evaluated th neurocognitive dysfunction between groups separated by the presence of IJVVI.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Akkawi NM, Agosti C, Borroni B, Rozzini L, Magoni M, Vignolo LA, Padovani A. Jugular valve incompetence: a study using air contrast ultrasonography on a general population. J Ultrasound Med. 2002 Jul;21(7):747-51. doi: 10.7863/jum.2002.21.7.747. PMID 12099562
- [Background] Silva MA, Deen KI, Fernando DJ, Sheriffdeen AH. The internal jugular vein valve may have a significant role in the prevention of venous reflux: evidence from live and cadaveric human subjects. Clin Physiol Funct Imaging. 2002 May;22(3):202-5. doi: 10.1046/j.1475-097x.2002.00418.x. PMID 12076346
- [Background] Dresser LP, McKinney WM. Anatomic and pathophysiologic studies of the human internal jugular valve. Am J Surg. 1987 Aug;154(2):220-4. doi: 10.1016/0002-9610(87)90185-1. PMID 3631396
- [Background] Sander D, Winbeck K, Etgen T, Knapp R, Klingelhofer J, Conrad B. Disturbance of venous flow patterns in patients with transient global amnesia. Lancet. 2000 Dec 9;356(9246):1982-4. doi: 10.1016/S0140-6736(00)03313-4. PMID 11130530
- [Background] Nedelmann M, Eicke BM, Dieterich M. Increased incidence of jugular valve insufficiency in patients with transient global amnesia. J Neurol. 2005 Dec;252(12):1482-6. doi: 10.1007/s00415-005-0894-9. Epub 2005 Jul 7. PMID 15999232
- [Background] Maalikjy Akkawi N, Agosti C, Anzola GP, Borroni B, Magoni M, Pezzini A, Rozzini L, Vignolo LA, Padovani A. Transient global amnesia: a clinical and sonographic study. Eur Neurol. 2003;49(2):67-71. doi: 10.1159/000068501. PMID 12584412